CLINICAL TRIAL: NCT04890054
Title: Screening More Patients for CRC Through Adapting and Refining Targeted Evidence-Based Interventions in Rural Settings (SMARTER CRC)
Brief Title: Screening More Patients for Colorectal Cancer Through Adapting and Refining Targeted Evidence-Based Interventions in Rural Settings, SMARTER CRC
Acronym: SMARTER CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Melinda Davis, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00020681; NCI-2021-01032 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020681 (Other: OHSU Knight Cancer Institute); UH3CA244298 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic; Patient Navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMARTER CRC Intervention Year 1 (Active Comparator): In year 1, patients receive mailed FITs from CCO, screening reminders from clinics, and patient navigation as appropriate; Health record data collected.
  Interventions: Other: Fecal Immunochemical Test; Other: Interview; Behavioral: Patient Navigation
- SMARTER CRC Usual Care (No Intervention): Usual clinical care

INTERVENTIONS:
Other: Fecal Immunochemical Test — Patients due for CRC screening are mailed a FIT test by the clinic or health plan
  Other Names: FIT; iFOBT; immunoassay fecal occult blood test; immunochemical fecal occult blood test; Immunochemical FOBT; immunologic fecal occult blood test
  Arms: SMARTER CRC Intervention Year 1
Other: Interview — Participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations
  Arms: SMARTER CRC Intervention Year 1
Behavioral: Patient Navigation — Clinic staff are trained in Navigation, patients with an abnormal FIT are contacted about colonoscopy by patient navigators
  Other Names: Patient Navigator Program
  Arms: SMARTER CRC Intervention Year 1

SUMMARY:
This study collects information to provide a model for how to rapidly adapt and scale-up multilevel interventions through clinic-health plan partnerships to reduce the burden of colorectal cancer (CRC) on the United states population. This study may improve colorectal cancer screening rates, follow-up colonoscopy, and referral to care in rural Medicaid patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Adapt, pilot, then test the implementation and scale-up of targeted direct mail and patient navigation programs.

OUTLINE:

This is an implementation-effectiveness trial of direct mail outreach and patient navigation intervention to improve rates of CRC screening. Eligible patients will be mailed a fecal immunochemical test (FIT). The mailed FIT and patient navigation interventions are a part of standard care and are carried out by the Medicaid health plan or clinic. Outcomes are tracked using reports from direct mail vendors, claims data from participating Medicaid health plans, clinic data from the electronic health record, chart review, and data from a REDCap database. The hypotheses will be tested using a two-arm cluster randomized trial design. Participating clinics will be randomized into two groups: Intervention and Usual Care. Medicaid health plans/ Coordinated care organizations (CCO) and clinic leadership participate in interviews and complete surveys.

The primary effectiveness outcome of this study is CRC screening likelihood in eligible Medicaid patients in intervention and control clinics at 6 months. Data will be collected at 6 time points: baseline, 6-months, 12-months, 18-months, 24-months, and 36-months.

Implementation outcomes and adaptations will be evaluated through interviews with clinic staff, patients, and CCO partners. Clinic staff in various roles related to the program (e.g., outreach workers, patient navigators, quality improvement leads) complete surveys and participate in interviews and observations at baseline, 6-9 months (post-implementation) and at approximately 12 months later, to assess clinic/health system level factors that may influence outcomes. Patients participate in interviews to explore patient experiences with the program. Regional and Organizational partners: CCO leaders, endoscopy providers (e.g., gastrointestinal specialists, general surgeons, primary care clinicians), and community organizations also participate in interviews.

ELIGIBILITY:
Inclusion Criteria:

* CCOs/CCO STAFF: Serving a majority of counties that are predominantly rural based on 2010 Rural-Urban Commuting Area (RUCA) codes (codes 4-10)
* CCOs/CCO STAFF: Willing to participate in data collection activities (e.g., producing claims data, interviews)
* CLINICS: Clinics will be eligible for the cluster randomization if there are 30 or more patients eligible for screening
* CLINICS: Are classified as rural according to RUCA (Codes 4-10) or Oregon Office of Rural Health designations
* CLINICS: Are served by CCOs agreeing to participate in the project
* CLINICS: Willing to implement the intervention into their clinic for the study
* CLINIC STAFF/PROVIDERS: Employed as a clinician or ancillary staff member in a participating clinic
* CLINIC STAFF/PROVIDERS: Willing to participate in data collection activities (e.g., interviews, observation, surveys)
* PATIENTS: Attributed to participating clinic
* PATIENTS: Are enrolled in Medicaid or dual eligible
* PATIENTS: Eligible for colorectal cancer (CRC) screening
* PATIENTS: For the subset of patients that will be invited to participate in key informant interviews, a 5th eligibility criteria is consented to participate
* COMMUNITY OR REGIONAL/ORGANIZATIONAL PARTNERS: (Includes endoscopy providers, community-based outreach workers, or leaders from regional or national organizations who participate in the pilot, pragmatic trial, or scale-up study)
* COMMUNITY OR REGIONAL/ORGANIZATIONAL PARTNERS: Involved in study activities (training, care delivery)
* COMMUNITY OR REGIONAL/ORGANIZATIONAL PARTNERS: Willing to participate in data collection activities (e.g., trainings, interviews, surveys)
* Elderly - Yes - we anticipate that a limited number of clinic and CCO staff, or community organization representatives may be elderly; we limit our patient recruitment to those aged 45-75
* Rural - Yes
* Inner city - No
* Low income - Yes
* Disabled - Yes
* Chronic care - Yes
* End of life - Yes - This is possible, but we predict limited numbers because of the types of individuals we are recruiting: clinic and CCO staff, and patients who are not currently in hospice care
* Minorities - Yes

Exclusion Criteria:

* CLINICS: Clinics are excluded if they have current or ongoing participating in other mailed fecal testing research projects in the Medicaid population
* PATIENTS: Are current for screening
* PATIENTS: Comorbid conditions that make patients poor candidates for screening based on clinical judgment (e.g., end-stage renal disease, enrollment in hospice)
* PATIENTS: Are not an established patient or for other reasons documented by the clinics
* All patients that we recruit will be at least 45 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5696 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Davis, PhD, Principal Investigator — OHSU Knight Cancer Institute; Gloria Coronado, PhD, Principal Investigator — University of Arizona
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-identifiable data is going to be available through the ACCSIS coordinating center as a public common data set across all the ACCSIS studies along with paper-specific de-identified data sets.
Time Frame: Available Now
URL: https://healthcaredelivery.cancer.gov/accsis/datashare

REFERENCES:
- [Derived] Coronado GD, Petrik AF, Leo MC, Coury J, Durr R, Badicke B, Thompson JH, Edelmann AC, Davis MM. Mailed Outreach and Patient Navigation for Colorectal Cancer Screening Among Rural Medicaid Enrollees: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e250928. doi: 10.1001/jamanetworkopen.2025.0928. PMID 40094661
- [Derived] Coury J, Coronado G, Currier JJ, Kenzie ES, Petrik AF, Badicke B, Myers E, Davis MM. Methods for scaling up an outreach intervention to increase colorectal cancer screening rates in rural areas. Implement Sci Commun. 2024 Jan 8;5(1):6. doi: 10.1186/s43058-023-00540-1. PMID 38191536
- [Derived] Coronado GD, Leo MC, Ramsey K, Coury J, Petrik AF, Patzel M, Kenzie ES, Thompson JH, Brodt E, Mummadi R, Elder N, Davis MM. Mailed fecal testing and patient navigation versus usual care to improve rates of colorectal cancer screening and follow-up colonoscopy in rural Medicaid enrollees: a cluster-randomized controlled trial. Implement Sci Commun. 2022 Apr 13;3(1):42. doi: 10.1186/s43058-022-00285-3. PMID 35418107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited clinics affiliated with three Medicaid health plans that serve rural counties in Oregon. Clinics had at least 30 age-eligible Medicaid or dually enrolled in Medicaid and Medicare; had CRC screening rates of 60% or lower; and operated in a geographic region designated as rural or frontier. Eligible individuals are ages 50-74 and eligible for CRC screening. Recruitment of clinics happened between May 2020-April 2021.
Pre-assignment Details: Stratified allocation assignments by clinic unit affiliation (hospital-affiliated, health care network-affiliated, clinic, etc.)
Units Other Than Participants: Clinics
Groups:
- SMARTER CRC Intervention Year 1: In year 1, patients receive mailed FITs from CCO, screening reminders from clinics, and patient navigation as appropriate; Health record data collected.
  Fecal Immunochemical Test: Patients due for CRC screening are mailed a FIT test by the clinic or health plan
  Interview: Clinic staff participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations
  Patient Navigation: Clinic staff are trained in Navigation, patients with an abnormal FIT are contacted about colonoscopy by patient navigators
- SMARTER CRC Usual Care: Patients receive usual clinical care in the SMARTER CRC clinics for people eligible for CRC screening.
  Interview: Clinic staff participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations.
Period: Overall Study
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care
Started | 2655; 14 Clinics | 3041; 14 Clinics
Patients | 2613; 14 Clinics | 3001; 14 Clinics
Staff | 42; 14 Clinics | 40; 14 Clinics
Completed | 2453; 14 Clinics (One clinic closed after randomization and before the intervention began. All staff completed research data collection activities.) | 2822; 14 Clinics
Not Completed | 202; 0 Clinics | 219; 0 Clinics
Not completed — Lost to Follow-up | 202 | 219

BASELINE CHARACTERISTICS:
Population: Patients of participating clinics included only. Demographics were not collect on staff participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care | Total
Number analyzed (Participants) | 2613 | 3001 | 5614
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (5.4) | 58.3 (5.6) | 58.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1334 | 1614 | 2948
  Male | 1279 | 1387 | 2666
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 190 | 325
  Not Hispanic or Latino | 2357 | 2583 | 4940
  Unknown or Not Reported | 121 | 228 | 349
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 97 | 50 | 147
  Asian | 30 | 21 | 51
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 16 | 19 | 35
  White | 1745 | 2029 | 3774
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 721 | 879 | 1600
Region of Enrollment [Number; unit: participants]
  United States | 2613 | 3001 | 5614
Insurance Status [Count of Participants; unit: Participants]
  Medicaid | 2157 | 2398 | 4555
  Dual Eligible | 456 | 603 | 1059
Rurality (RUCA Codes) [Count of Participants; unit: Participants]
  Metropolitan | 70 | 730 | 800
  Micropolitan | 1722 | 1680 | 3402
  Small Town | 431 | 156 | 587
  Rural | 384 | 432 | 816
  Unknown or Missing | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Likelihood of Any Colorectal Cancer (CRC) Screening (for Study-eligible Patients)
Description: Adjusted 6-month any CRC screening for enrollees in clinic units. These values are predicted estimates rather than crude number [%] generated using marginal standardization and accounting for clustering and covariates (i.e., sex, age, and Medicaid health plan). Claims and vendor data were used to determine whether or not the patient completed CRC screening (i.e., fecal testing, FIT-DNA, sigmoidoscopy, CT colonography, or colonoscopy). To assess effectiveness of CRC screening completion, we used the generalized form of hierarchical linear model (binomial distribution with logit link) to account for clustering of patients within clinics and the assignment to arm at the clinic level.
Time Frame: Primary outcome at 6 months following CCO eligible patient list pull date,
Population: Intention to treat, multi-level within clinics. One clinic closed immediately after randomization and before patients could be determined eligible before the intervention began.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Groups:
- SMARTER CRC Intervention Year 1: In year 1, patients receive mailed FITs from CCO, screening reminders from clinics, and patient navigation as appropriate; Health record data collected.
  Fecal Immunochemical Test: Patients due for CRC screening are mailed a FIT test by the clinic or health plan.
  Interview: Clinic staff participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations.
  Patient Navigation: Clinic staff are trained in Navigation, patients with an abnormal FIT are contacted about colonoscopy by patient navigators.
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care
Number analyzed (Participants) | 2613 | 3001
Percentage of participants | 11.8 [10 to 13.5] | 4.5 [3.6 to 5.4]

2. Secondary Outcome: Completion of CRC Screening
Description: Completed CRC screening at 12 months. Claims and vendor data were used to determine whether or not the patient completed CRC screening (i.e., fecal testing, FIT-DNA, sigmoidoscopy, CT colonography, or colonoscopy).
Time Frame: Up to 12 months
Population: Intent to treat, multi-level within clinics. One clinic closed after randomization and before the intervention began.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care
Number analyzed (Participants) | 2613 | 3001
Percentage of participants | 16.8 [15.3 to 18.2] | 9 [8.0 to 10.0]

3. Secondary Outcome: Rate of CRC Screening Among the Intervention-eligible Population
Description: In the intervention clinics only, the list of patients eligible for screening was scrubbed by clinics. This percent is the N completed CRC screening out of the N included in intervention outreach after clinics scrubbed the list of eligible patients.
Time Frame: 6 months
Population: Patients NOT excluded during the clinic scrub, expected for intervention components.
Measure: Count of Participants; unit: Participants
Arm/Group | SMARTER CRC Intervention Year 1
Number analyzed (Participants) | 2613
Participants | 181

4. Secondary Outcome: Time to Screening From Study-eligible Patient List Pull
Description: Days from study-eligible patient list pull to abnormal FIT result. Number of days at individual level.
Time Frame: Up to 12 months
Population: Intent to treat eligible patients at clinics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care
Number analyzed (Participants) | 2613 | 3001
Days | 118.5 (293.9) | 103.2 (383.2)

5. Secondary Outcome: Abnormal FIT Results
Description: Number of participants with abnormal FIT Results
Time Frame: 6 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: Patients receive usual clinical care in the SMARTER CRC clinics for people eligible for CRC screening.
  Interview: Clinic staff participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations.
Arm/Group | SMARTER CRC Intervention Year 1 | Usual Care
Number analyzed (Participants) | 2613 | 3001
Participants | 19 | 7

6. Secondary Outcome: Patient Navigation Trainings (Intervention Group)
Description: Clinic participation (i.e., attendance) in patient navigation training, Year 1 clinical trial
Time Frame: Up to 12 months
Population: A subset of the total population of clinic staff, who were invited to the patient navigation training
Measure: Count of Participants; unit: Participants
Arm/Group | SMARTER CRC Intervention Year 1
Number analyzed (Participants) | 42
Participants | 22

7. Secondary Outcome: Patient Navigation Completed (Intervention Group)
Description: Patient navigation implemented = one or more live phone contact with the patient (binary at the individual level).
Time Frame: Up to 12 months
Population: Patients in intervention clinics eligible for navigation to colonoscopy due to FIT test result or medical factors
Measure: Count of Participants; unit: Participants
Arm/Group | SMARTER CRC Intervention Year 1
Number analyzed (Participants) | 35
Participants | 22

8. Secondary Outcome: Follow-up Colonoscopy Completion
Description: The percentage of patients with abnormal FIT who completed follow-up colonoscopy within 12 months
Time Frame: Up to 12 months
Population: Intention to treat, patients in clinics
Measure: Number; unit: Percent of participants
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care
Number analyzed (Participants) | 2613 | 3001
Percent of participants | 49.1 | 19.7

9. Secondary Outcome: Time to Colonoscopy From Abnormal FIT Result
Description: Days from abnormal FIT result to completion of follow-up colonoscopy. Number of days at the individual level.
Time Frame: Up to 12 months
Population: Intention to treat, patients in clinics
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | SMARTER CRC Intervention Year 1 | SMARTER CRC Usual Care
Number analyzed (Participants) | 2613 | 3001
Days | 96.3 [72.6 to 119.9] | 114.6 [50.0 to 179.2]

10. Secondary Outcome: Adenomas or Cancers Detected
Description: Whether or not eligible patient had an adenoma or cancer detected. Binary at individual level.
Time Frame: Up to 12 months
Population: Intention to treat, patients in clinics
Measure: Number; unit: participants
Arm/Group | SMARTER CRC Intervention Year 1 | Usual Care
Number analyzed (Participants) | 2613 | 3001
participants
  Adenomas | 7 | 14
  Cancers | 1 | 4

11. Secondary Outcome: Key Implementation Barriers
Description: Qualitative key informant interviews with clinic and payer stakeholders to identify implementation barriers.
Time Frame: Up to 36 months
Population: Clinic or CCO staff, including patient navigators, who were involved in implementation of the intervention
Measure: Count of Participants; unit: Participants
Groups:
- SMARTER CRC Intervention and Usual Care Year 1: Clinic staff from both the intervention and usual care groups participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations.
Arm/Group | SMARTER CRC Intervention and Usual Care Year 1
Number analyzed (Participants) | 82
Participants
  COVID disruptions | 4
  Staffing Disruptions | 19
  Mailing Delays | 5
  Did Not Mention | 54

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the course of 2 years.
Groups:
- SMARTER CRC Intervention Patients: In year 1, patients receive mailed FITs from CCO, screening reminders from clinics, and patient navigation as appropriate; Health record data collected.
  Fecal Immunochemical Test: Patients due for CRC screening are mailed a FIT test by the clinic or health plan.
- Usual Care Patients: Patients receive usual clinical care in the SMARTER CRC clinics for people eligible for CRC screening.
  Interview: Clinic staff participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations.
- Intervention Staff Members: Clinic staff participate in interviews to evaluate the implementation of the mailed FIT and patient navigation programs by the clinics and regional organizations. They also receive patient navigation training.
- Usual Care Staff Members: Clinic staff participate in interviews to evaluate outcomes in the usual care group.
Arm/Group | SMARTER CRC Intervention Patients | Usual Care Patients | Intervention Staff Members | Usual Care Staff Members
All-Cause Mortality (participants affected / at risk) | 0/2613 | 0/3001 | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/2613 | 0/3001 | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/2613 | 0/3001 | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT04890054/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04890054/ICF_001.pdf